CLINICAL TRIAL: NCT00446927
Title: SPY Imaging System: Its Role in Pediatric Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Brian Kogon, Associate professor, surgery, Emory University
Other Study IDs: IRB00001298
Record Dates: First submitted 2007-03-08; First posted 2007-03-13 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Cardiopulmonary Bypass; Congenital Heart Defects
Keywords: Pediatrics; Cardiology; Cardiopulmonary Bypass; Heart Surgery; Cardiac Catheterization; Echocardiography; Imaging; ICG green dye
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The current method of evaluating the surgical repair during surgery is limited to echocardiography (a noninvasive diagnostic procedure that uses ultrasound to study the structure and motions of the heart) or an invasive procedure called cardiac catheterization.

The SPY imaging system makes use of the fluorescence properties of indocyanine green (ICG) to obtain high quality images in blood vessels. ICG is a green dye used to test heart output. The use of the SPY imaging system during surgery may provide valuable information regarding successful vessel connection and the area remaining unblocked.

This study will compare the results of images to echocardiography and conventional angiography results.

With SPY imaging, congenital heart surgeons would be able to check the quality of the procedure and revise, redo or perform additional procedures as dictated by the images before the patient leaves the operating room.

DETAILED DESCRIPTION:
It would be advantageous to detect potential problems with vessel and anastomotic patency prior to leaving the operating room. The SPY imaging system makes use of the fluorescence properties of Indocyanine Green (ICG) to obtain high quality images of blood vessels. Unlike conventional angiography, indocyanine green fluorescence imaging offers the potential for a reliable, non invasive, inexpensive and rapid method of intraoperative assessment of vessel and anastomotic patency.

This type of imaging resource could be invaluable in a repair such as:

1. coronary artery re-implantation following arterial switch procedure for transposition of the great arteries, anomalous coronary artery from the pulmonary artery repair, or aortic root replacement,
2. coarctation of the aorta,
3. Blalock-Taussig shunt, right-ventricle-to-pulmonary artery shunt, or cavopulmonary connection for single ventricle palliation, and
4. branch or distal pulmonary artery reconstruction/unifocalization in tetralogy of Fallot and pulmonary atresia/ventricular septal defect.

The SPY imaging system is feasible for a variety of congenital heart defects and can provide valuable information regarding vessel and anastomotic patency.

Specific Aim 1: Evaluate quality of images for clarity and ability to visualize desired anatomic area

Specific Aim 2: Compare results of images to echocardiography and conventional angiography results

* Part 1. Compare the results of pre-repair intra-operative SPY images to preoperative echocardiography results, and cardiac catheterization results when available
* Part 2. Compare the results of post-repair intraoperative SPY images to postoperative echocardiography results, and cardiac catheterization results when available

Approximately 40 patients in total will be enrolled in the study - 10 who have undergone coronary reimplantation, 10 who have undergone repair of coarctation of the aorta, 10 who have undergone a palliative shunting procedure, and 10 who have undergone pulmonary artery reconstruction.

Echocardiography:

Preoperative, intraoperative, and postoperative cardiac catheterization reports will be analyzed.

Cardiac catheterization:

Preoperative and postoperative cardiac catheterization reports will be analyzed.

SPY imaging:

ICG green will be administered in the following doses: 1.25 mg in infants (< 1 year), 2.5 mg in children (<16 years), and 5 mg in adult size patients (17-18 years of age). Doses will be injected in 1 ml volumes directly into the aorta, right ventricle or pulmonary artery, depending upon the procedure. Repeat dosing and imaging may be performed if needed. The total dose of dye will be limited to 2 mg/kg. Images will be obtained in the operating room prior to commencing and after weaning from cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing congenital heart operations at Children's Healthcare of Atlanta.
* Less than or equal to 18 years of age.
* Arterial switch procedure
* Anomalous coronary artery from the pulmonary artery repair
* Aortic root replacement
* Coarctation of the aorta repair
* Blalock-Taussig shunt
* Right ventricle-to-pulmonary artery shunt
* Cavopulmonary shunt
* Branch or distal pulmonary artery reconstruction
* Unifocalization of aortopulmonary collaterals

Exclusion Criteria:

* Known sensitivity to ICG, iodides or shellfish
* Inability to obtain informed consent
* > 18 years of age

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study patients will be consented in the pre-operative clinic, Cardiac Intesive Care unit or from the Cardiac Step-down Unit.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kogon, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Bonhoeffer P, Bonnet D, Piechaud JF, Stumper O, Aggoun Y, Villain E, Kachaner J, Sidi D. Coronary artery obstruction after the arterial switch operation for transposition of the great arteries in newborns. J Am Coll Cardiol. 1997 Jan;29(1):202-6. doi: 10.1016/s0735-1097(96)00433-0. PMID 8996315
- [Background] Tanel RE, Wernovsky G, Landzberg MJ, Perry SB, Burke RP. Coronary artery abnormalities detected at cardiac catheterization following the arterial switch operation for transposition of the great arteries. Am J Cardiol. 1995 Jul 15;76(3):153-7. doi: 10.1016/s0002-9149(99)80048-4. PMID 7611150
- [Background] Bonnet D, Bonhoeffer P, Piechaud JF, Aggoun Y, Sidi D, Planche C, Kachaner J. Long-term fate of the coronary arteries after the arterial switch operation in newborns with transposition of the great arteries. Heart. 1996 Sep;76(3):274-9. doi: 10.1136/hrt.76.3.274. PMID 8868989
- [Background] Ibarra-Perez C, Castaneda AR, Varco RL, Lillehei CW. Recoarctation of the aorta. Nineteen year clinical experience. Am J Cardiol. 1969 Jun;23(6):778-84. doi: 10.1016/0002-9149(69)90371-3. No abstract available. PMID 5785157
- [Background] Parsons CG, Astley R. Recurrence of aortic coarctation after operation in childhood. Br Med J. 1966 Mar 5;1(5487):573-7. doi: 10.1136/bmj.1.5487.573. No abstract available. PMID 5908418
- See also: Click here for more information about the SPY Imaging System — http://www.novadaq.com/